CLINICAL TRIAL: NCT07168629
Title: A Community Health Worker Intervention to Improve Lung Cancer Screening Uptake in Community Health Centers
Acronym: CHATS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Eduardo, Assistant Professor Departments of Medicine and Healthcare Delivery and Population Sciences, Baystate Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2151088-4; 1K08CA289097-01 (NIH)
Record Dates: First submitted 2025-08-13; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer; Tobacco Use
Keywords: lung cancer screening; tobacco treatment; community health workers; community health centers
MeSH Terms: conditions — Lung Neoplasms; Tobacco Use

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (Active Comparator): Will receive educational materials about lung cancer screening and tobacco treatment.
  Interventions: Other: Enhanced Usual Care
- Intervention (Experimental): Will receive a four-part community health worker-delivered intervention to improve LCS uptake, which includes: 1) patient outreach, 2) patient-centered shared decision-making, 3) smoking cessation counseling, and 4) navigation of logistical barriers
  Interventions: Behavioral: Community health worker delivered outreach, shared decision-making, tobacco treatment, and navigation

INTERVENTIONS:
Behavioral: Community health worker delivered outreach, shared decision-making, tobacco treatment, and navigation — The CHW will perform: 1) patient outreach 2) patient-centered shared-decision making, 3) smoking cessation counseling, and 4) navigation of logistical barriers
  Arms: Intervention
Other: Enhanced Usual Care — After randomization, the control group will receive the same mailed LCS educational materials as the intervention group and encouraged to discuss screening with their PCP, the typical pathway through which patients enter the LCS program.
  Arms: Enhanced Usual Care

SUMMARY:
Lung cancer screening (LCS) can reduce lung cancer-related mortality by 20%, but only 5-10% of eligible individuals have received an initial LCS. The goal of this study is to partner with community stakeholders to jointly develop and pilot test a multi-component community health worker-delivered intervention targeting key barriers to improve LCS and tobacco treatment utilization. The proposed activities will lay the groundwork for a subsequent R01 grant, conducting a fully powered randomized clinical trial to establish CHWs as an evidence-based practice that will facilitate access to screening and tobacco treatment, to reduce lung cancer mortality.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death, and lung cancer screening (LCS) can reduce lung cancer-related mortality by 20%. However, only 5-10% of eligible individuals have received an initial LCS exam. Community health worker (CHW) interventions have been effective at promoting screening in other cancer settings. Whether a CHW-delivered intervention can be effective in the context of LCS and address key barriers to receiving LCS remains unknown. The goal of this study is to develop and pilot test a four-part CHW-delivered intervention to improve LCS uptake, which includes: 1) patient outreach, 2) patient-centered shared decision-making, 3) smoking cessation counseling, and 4) navigation of logistical barriers. Our central hypothesis, based on our qualitative work and informed by the expanded Health Belief Model, proposes that a CHW-delivered intervention can address key modifiable factors to improve LCS awareness, engagement, and barriers to accessing care, leading to increased LCS uptake. Our aims are to: Jointly "transcreate" a CHW-delivered intervention to increase LCS uptake among patients served by community health centers (Aim 1); conduct a pilot randomized controlled trial of the intervention (Aim 2a); and obtain empiric estimates of effect size in LCS and tobacco treatment utilization (Aim 2b). We first seek to jointly "transcreate" the intervention with our community advisory board, comprised of key stakeholders in LCS and patients with lived experience, applying the Transcreation Framework for Community-Engaged Behavioral Interventions. Then we will conduct a pilot randomized controlled trial of the CHW-delivered intervention at Baystate Health's three community health centers. We will randomize 80 LCS-eligible individuals (40 in each arm) to either the intervention or enhanced usual care (i.e., mailed LCS educational materials and usual LCS as per primary care provider). Primary pilot outcomes are focused on feasibility, including participant recruitment, measure completion, retention, fidelity, and acceptability. We will also conduct an evaluation of secondary trial outcomes, including LCS and tobacco treatment utilization, as well as explore potential mediators (e.g., knowledge, facilitation of logistical barriers). The proposed activities will provide me with crucial skills in community-engaged research, implementation science, and clinical trial design, and launch my career as a clinician-scientist dedicated to addressing lung cancer mortality. This work will also lay the groundwork for a subsequent R01 grant conducting a fully powered randomized controlled trial of the CHW-delivered intervention that directly addresses top priorities from the President's Cancer Moonshot and NCI's mission to develop multi-level interventions that facilitate access to cancer screening and reduce lung cancer mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the age of 50 and 80.
* Potentially eligible for LCS according to the Electronic Health Record smoking history.
* Receive their primary care at Mason Square, High Street, or Brightwood community health centers.
* English- or Spanish- speaking.

Exclusion Criteria:

* Not eligible for lung cancer screening based on age (age < 50 or > 80 years) or smoking history (has not smoked more than 20 pack-years of tobacco cigarettes or quit more than 15 years ago).
* Have received a lung cancer screen in the past.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Feasiblity | once a month until study trial ends, an average one year
  Recruitment & enrollment: # of participants approached, met eligibility, and randomized Baseline Measures (see Table 5): Completeness of data collection. Retention: Loss of follow-up, reason for discontinuation, completeness of post-intervention data
Fidelity | once a month until study trial ends, an average of 1 year
  Duration of SDM and Smoking cessation Navigation: amount of time spent per call
Fidelity | once a month until study trial ends, an average of 1 year
  Completion of SDM and Smoking Cessation
  SDM OPTION Scale: measures 12 SDM items on a 5-point scale with response values ranging from "not observed" (value of 0) to "exhibited at a very high standard" (value of 4), with a total possible score ranging from 0 to 48.
  CMS SDM elements: reduced lung cancer mortality, false positive, overdiagnosis, radiation exposure, annual screening, smoking cessation, follow-up testing, and diagnostic procedures.
Fidelity | once a month until study trial ends, an average of 1 year
  SDM aid use and resources utilized
Fidelity | once a month until study trial ends, an average of 1 year
  Referral to tobacco treatment services and type of referral (e.g., telephone quit line, in-person), nicotine replacement therapy.
Acceptability | 3 months post enrollment (for study participant) and through study completion, an average of 1 year (for CHW staff)
  CHWs: Encounter logs documenting participant concerns and barriers to LCS
  Qualitative Interviews:
  Participants (N=15): Completed at the 3-month follow-up in a private setting, duration ~40-45 minutes, to assess the overall experience with the CHW intervention and barriers to LCS.
  CHWs (N=3): One 45-minute interview with each CHW after completing their last intervention delivery during the trial period.

SECONDARY OUTCOMES:
LCS referral | 3 months post study enrollment
  Referral for LCS: Order either by CHW or PCP referring participant to LCS program.
LCS uptake | Baseline and post intervention, 3 months post study enrollment
  Receipt of LCS pre and post intervention
Tobacco Treatment receipt | 3 months post study enrollment
  Receipt of tobacco treatment: initiation and type of treatment
Tobacco Treatment Duration | 3 months post study enrollment
  Duration of tobacco treatment and cessation attempts.
Tobacco Cessation | 3 months post study enrollment
  Tobacco Cessation: # of quit attempts

OTHER OUTCOMES:
LCS knowledge | Baseline and at 3 months post-enrollment
  LCS knowledge LCS-12: 12-item instrument measuring LCS knowledge, indications for screening and potential risks
LCS beliefs and barriers | At baseline and at 3 months post-enrollment
  LCS Health Belief Scale: 35-item instrument based on the Expanded Health Belief Model that measures perceived risk of lung cancer (3 items), knowledge and perceived LCS benefits (6 items), perceived LCS barriers (17 items), and self-efficacy (9 items; e.g. patient confidence in ability to arrange and complete LCS). Item responses use a 4-point Likert scale (e.g. strongly agree to strongly disagree).
Trust in Navigator | 3 months post-enrollment
  Trust in Navigator Scale: 6-item instrument developed to measure interpersonal trust in a patient's navigator (i.e., the CHW), adapted from the trust in physician scale.
Values-based SDM | 3 months post-enrollment
  SDM Process Survey: 4-item scale that measures whether the conversation discussed harms and benefits, and decisional preferences.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Pacheco, Study Director — Baystate Health

IPD SHARING:
Plan to Share IPD: No
Sharing qualitative data such as transcriptions from interviews can potentially reveal sensitive information and identify individual participants. The higher level of redaction needed to remove potentially-identifying and sensitive information would substantially reduce the utility of transcripts in future analyses.To ensure this group's participation and honest responses, we will not share transcripts or coding summaries from participant or community health worker interviews.
  The goal of this pilot trial is to provide preliminary information to support a future fully powered randomized trial to address disparities in lung cancer in Black and Hispanic communities. Given that these community members have historically been subject to unethical research practices, we will limit the potential for further distrust by not sharing de-identified information outside of the study team or its collaborators.